CLINICAL TRIAL: NCT02539589
Title: Evaluation of Becoming a Responsible Teen (BART)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5 TP1AH000003-02-00 BART
Record Dates: First submitted 2015-08-28; First posted 2015-09-03 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Becoming a Responsible Teen (BART) (Experimental): Becoming a Responsible Teen (BART) is the treatment condition. BART is an out of school educational program that intends to provide cognitive behavioral training to reduce HIV risk.
  Interventions: Behavioral: BART
- Healthy Living (Active Comparator): Healthy Living is the control counterfactual condition. It is a knowledge-based intervention that aims to impact nutrition, healthy eating, body image, and exercise.
  Interventions: Behavioral: Healthy Living

INTERVENTIONS:
Behavioral: BART — BART is an out of school educational program that intends to provide cognitive behavioral training to reduce HIV risk. It is intended to be implemented in 8 sessions lasting 1.5-2 hours. Sessions are to be implemented by a male and female health educator in small gender specific groups of 5-15 participants.
  Arms: Becoming a Responsible Teen (BART)
Behavioral: Healthy Living — Healthy Living is a knowledge-based intervention that intends to provide one HIV information-only session and seven sessions on nutrition, healthy eating, body image, and exercise. It is intended to be implemented in 8 sessions lasting 1.5-2 hours. Sessions are to be implemented by a male and female health educator in small gender specific groups of 5-15 participants.
  Arms: Healthy Living

SUMMARY:
The purpose of the study is to determine the impact of the offer to participate in Becoming a Responsible Teen (BART) (treatment) relative to the offer to participate in Healthy Living (control) on two self-reported sexual behaviors (condom use and frequency of sex) six months after the end of treatment.

DETAILED DESCRIPTION:
The Policy & Research Group (PRG) will be evaluating the Becoming a Responsible Teen (BART) curriculum. As part of the program, participants will be randomly assigned to receive either BART (treatment) or the Healthy Living (control) curriculum. BART is an eight-session group-level HIV/AIDS risk reduction curriculum based on Social Learning Theory and Self-efficacy Theory. The Healthy Living curriculum consists of the first session of BART (HIV information-only) followed by seven sessions of nutrition and physical activity education. The study is an individual randomized controlled trial in which eligible, consenting participants were randomly assigned by evaluators to intervention or control conditions. Random assignment occurred after evaluation consent/assent had been obtained and before the provision of any programming or collection of baseline data. There was no difference in the consent process for the intervention or control groups. Most study participants were randomized at approximately the same time-the first day of programming. Others were randomized when they showed up to a study site for the first time sometime during the first or second week of programming. Participant assignment was blocked by employment site, work shift, and gender. Baseline, outcome, and covariate data were collected via self-administered questionnaires that were scheduled at the following times: baseline (before the first program session attended); immediate post-program follow-up; 6-month post-program follow-up; and 12-month post-program follow-up. The study took place in New Orleans, Louisiana, as part of an educational component of a summer employment program funded by the city government. The government program contracts with multiple local community-based organizations (CBOs) to offer summer camps, internships, job training, and employment opportunities for youth ages 14 to 21 who reside in Orleans Parish. Each summer, these CBOs implemented the BART and Healthy Living programs as a component of their summer programming. Youth were recruited and enrolled during three consecutive summers (2012 to 2014), with programming ending each summer by late July. Six-month follow-up data collections occurred February to July of each year. Twelve-month follow-up data collections were generally offered from July to January of each year.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14-18
* City youth worker assigned to a job site that is offering program
* Provide parental consent (if under age 18) and participant assent to participate in the study.

Exclusion Criteria:

* Not have previously participated in any of the following pregnancy/HIV prevention programs:

  * 4 Real Health
  * Becoming a Responsible Teen (BART)
  * Healthy Living
  * Staying Mature and Responsible Towards Sex (SMARTS)
  * Sisters Informing Healthy Living and Empowering (SIHLE)
  * Project AIM
  * Making Proud Choices
  * Be Proud Be Responsible, or
  * Focus on Your Future

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 850 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Two questionnaire items measuring consistency of condom use | 6 months after the end of intervention
  The outcome is measured as the proportion of times in the past three months a person reports having any type of sex without using a condom. The outcome variable is calculated from the following items on the Questionnaire administered 6 months after the programs end:
  * In total, how many times have you had any type of sex in the past 3 months?
  * Now, think about the number of times that you had any type of sex in the past 3 months. How many of those times did you use condoms?
  The resulting variable is a continuous proportion with values that range from 0 to 1, where 0 indicates that a person has not engaged in sex without a condom in the past three months, and 1 indicates that the person has engaged in sex without a condom 100% of the times they had sex in the past three months.

SECONDARY OUTCOMES:
One questionnaire item measuring frequency of sexual activity | 6 months after end of intervention
  The outcome is measured as the number of times in the past three months a person reports having any type of sex
  The measure is taken directly from the following item on the Questionnaire:
  • In total, how many times have you had any type of sex in the past 3 months?
  The variable is continuous, with values ranging from 0 to k, where 0= no sexual activity reported in past 3 months and k = number of times sex reported.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenner, PhD, Principal Investigator — The Policy & Research Group

REFERENCES:
- [Background] Walsh S, Jenner E, Leger R, Broussard M. Effects of a Sexual Risk Reduction Program for African-American Adolescents on Social Cognitive Antecedents of Behavior Change. Am J Health Behav. 2015 Sep;39(5):610-22. doi: 10.5993/AJHB.39.5.3. PMID 26248171
- [Background] Demby H, Gregory A, Broussard M, Dickherber J, Atkins S, Jenner LW. Implementation lessons: the importance of assessing organizational "fit" and external factors when implementing evidence-based teen pregnancy prevention programs. J Adolesc Health. 2014 Mar;54(3 Suppl):S37-44. doi: 10.1016/j.jadohealth.2013.12.022. PMID 24560075